CLINICAL TRIAL: NCT02090374
Title: Development of Human Nasal Challenge Models With Microbial Constituents and Grass Pollen: Monophosphoryl lipidA, Poly-inosine-cytosine, Poly-inosine-cytosine Stabilised With Poly-L-lysine and Carboxymethylcellulose, Resiquimod, Tuberculin and Timothy Grass Pollen
Brief Title: Development of Human Nasal Challenge Models With Microbial Constituents and Grass Pollen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 13SM1837; P45058 (Other Grant/Funding Number: NIHR Imperial Biomedical Research Council Grant)
Record Dates: First submitted 2014-03-11; First posted 2014-03-18 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Allergic Rhinitis; Asthma; Latent Tuberculosis
Keywords: Allergy; Asthma; Biomarkers; Chemokines; Cytokines; Eosinophil; Gene Expression; Grass pollen; Hay Fever; Human Challenge Study; Inflammation; Innate Immune Response; Lipopolysaccharide; Mucosal Lining Fluid; Nasal; Nasorption; Respiratory; Respiratory Tract Infection; T cells; Tuberculosis; Virus
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Latent Tuberculosis; Hypersensitivity; Rhinitis, Allergic, Seasonal; Inflammation; Respiratory Tract Infections; Tuberculosis; Virus Diseases | interventions — poly ICLC; Poly I-C; resiquimod; PHLPVI protein, Phleum pratense; Vitamin D; Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Poly ICLC dose escalation (Experimental): Poly ICLC nasal challenge dose escalation 10ug, 100ug, 500ug
  Interventions: Other: Poly ICLC
- Poly ICLC highest dose (Experimental): Poly ICLC nasal challenge single dose of 1000ug
  Interventions: Other: Poly ICLC
- Poly I:C single dose (Experimental): Poly I:C nasal challenge single dose 500ug
  Interventions: Other: Poly I:C
- R848 high dose (Experimental): R848 nasal challenge 10ug
  Interventions: Other: R848
- R848 low dose (Experimental): R848 nasal challenge low dose 1-2ug (0.02ug/kg)
  Interventions: Other: R848
- Grass pollen (Experimental): Timothy grass pollen nasal challenge
  Interventions: Other: Timothy Grass Pollen
- Vitamin D supplementation (Experimental): Vitamin D 4000U orally daily
  Interventions: Other: Vitamin D
- Tuberculin (Experimental): Tuberculin PPD nasal challenge
  Interventions: Other: Tuberculin

INTERVENTIONS:
Other: Poly ICLC — Dose escalation: 10ug, 100ug, 500ug Highest dose: 1000ug
  Arms: Poly ICLC dose escalation; Poly ICLC highest dose
Other: Poly I:C — Single dose: 500ug
  Arms: Poly I:C single dose
Other: R848 — High dose: 10ug Low dose: 1-2ug
  Other Names: Resiquimod
  Arms: R848 high dose; R848 low dose
Other: Timothy Grass Pollen — Dose: 5000 SQ-U/100µl
  Arms: Grass pollen
Other: Vitamin D — 4000U orally
  Arms: Vitamin D supplementation
Other: Tuberculin — Tuberculin PPD
  Arms: Tuberculin

SUMMARY:
The investigators propose the development of a range of nasal spray challenge models to study the way the nose can respond to different types of nasal challenge that elicit different forms of inflammation.

The investigators will carry out nasal challenge with bacterial and viral components and allergens. In this way the nasal upper respiratory tract mucosa is challenged with stimuli of the immune system, causing various types of inflammation. Samples will be taken by blotting the nostril surface and by scraping off tiny surface samples.

The nose will be sprayed with a substance that is a single part of a bacteria or virus, or with an allergen. The material delivered by nasal spray is of high purity and is sterile, containing no live bacteria or viruses. The nasal spray substance contains molecular patterns that are recognised as foreign by the immune system, and at the right dose should stimulate the immune system, causing mild nasal inflammation. The study employs noninvasive methods of sampling using absorptive strips. These strips look and feel like tissue paper, and are applied to each nostril for a period of 1 min. A few pinhead-sized tissue samples are taken from inside the nose, using a small disposable sterile plastic probe that has a tiny scoop on its end. In the nasal lining fluid and tissue samples, measurement will taken of a range of molecules and cells that protect against infections and help the immune response.

By spraying the nose with a challenge agent in this manner, the nasal immune response can be assessed, which can help us better understand how the human immune system cells and molecules respond to bacteria and viruses. In the future, this may allow the testing of new drugs and vaccines, by seeing if they decrease or stop the inflammation after the nasal challenge.

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODOLOGY

The study involves 3 parts with different nasal spray challenges being administered to subjects:

1. Bacterial or viral components, comprising one of the following in a particular patient;

   1. MPLA (monophosphoryl lipid A) resembles bacterial lipopolysaccharide
   2. PolyIC (polyinosinic and cytidylic acids): viral component
   3. PolyICLC (polyIC stabilised with polyLlysine): viral component
   4. Resiquimod: viral mimic
2. Tuberculin: partially purified protein derivative (PPD) from Mycobacterium bovis, the bacteria that causes TB.
3. Allergen: The nasal spray challenge agent is Timothy grass pollen.

RECRUITMENT

The aim is to recruit a total of 174 subjects. Subjects will be identified through advertisements in the newspapers, posters on the campus, GP services, outpatients clinics at St. Mary's hospital including TB clinics at St. Mary's Hospital. We will gain fully informed consent. All data will be managed as per GCP and local Information Governance guidelines.

NUMBER OF SUBJECTS AND DOSING

PART 1: Nasal ascending dose challenge with microbial constituents using MPLA, polyIC, polyICLC and resiquimod. This is divided into part A and part B.

PART 1A (n=32): Incremental Ascending Dose Study based on Tolerability and SAM. 4 cohorts of 8 healthy volunteers (4 of 8 with allergies to grass pollen, house dust mite, or history of hay fever). One cohort for each microbial constituent. Each cohort will be given a nasal saline control challenge and three ascending doses of the nasal microbial constituent challenge:

* 10μg of microbial constituent in 100μl of saline
* 100μg of microbial constituent in 100μl of saline
* 500μg of microbial constituent in 100μl of saline

PART 1B (n=64): Single Top Dose with Additional Special Sampling Probe (SSP) and Curettage, Single Cohort of up to 16 Healthy Volunteers (8 of 16 allergies to grass pollen, housedust mite, history of hay fever). Each subject given saline control and single top dose after establishing tolerability & SAM response.

RESIQUIMOD:

Part B will see 10μg per nostril being given to 36 volunteers:

12 allergic asthmatics 12 atopic volunteers 12 non-atopic volunteers

PART 2: Nasal ascending dose challenge with tuberculin. This is divided into part A and part B.

PART 2A (n=16): This comprises a total of 16 latent TB (LTB) subjects,This group is subdivided into 4 cohorts of 4 subjects according to the dose of the tuberculin being administered;

* 0.1 TU in 100μl, n = 4
* 1.0 TU in 100μl, n = 4
* 2.0 TU in 100μl, n = 4
* 5.0 TU in 100μl, n = 4 Each cohort has only 1 challenge. The starting dose is very low at 0.1 TU. If it is well tolerated, the subject will proceed to the next higher dose of 1.0 TU. If this is also well tolerated, the subject will proceed to the next higher dose of 2.0 TU and then to the highest dose of 5.0 TU in this group ensuring the safety of subjects at all times.

PART 2B (N=16): Top dose with additional sampling. This comprises of 16 people in two groups (8 healthy volunteers and 8 subjects with latent TB).

Group 1: Latent TB subject, no. of people = 8 This group will receive the top dose (5-10.0 TU) of the tuberculin challenge. Out of the 8 subjects in each group, 2 will receive placebo (saline dummy spray) and the remaining 6 will be given the tuberculin spray challenge.

Group 2: Healthy volunteers, no. of people = 8 This group will also receive the top dose (5-10.0 TU) of the tuberculin challenge, subject to tolerability. Out of the 8 subjects, 2 will receive the placebo (saline dummy spray) and the remaining 6 will be given the tuberculin spray challenge

PART 3 (n=46): Nasal Allergen Challenge with Timothy Grass Pollen

Initially 30 people shall be studied: one group of 12 people have hay fever, one group of 12 people have asthma with grass pollen allergy, and a group of 6 people are nonallergic and do not have asthma. In an additional group,16 people with hay fever shall be studied by taking continuous samples of the surface nasal lining fluid using a special sampling probe (SSP) following the nasal spray challenge.

1. Group 1: people with hay fever, n = 12
2. Group 2: people with allergic asthma, n = 12
3. Group 3: healthy, nonatopic people, n = 6
4. Additional Group 4: people with hay fever, n=16

NASAL PROCEDURES IN THE STUDY

1. Nasal washing (nasal lavage): At the start of the day, nasal washings in the nose will be carried out by passing a small volume of salt water (saline) fluid into the nose. This procedure is carried out before other procedures to clean up the nose. The fluid obtained from the nasal washings is discarded and not analysed.
2. Nasal lining fluid absorption (nasosorption or SAM): A small strip of absorbent material, that looks and feels like soft tissue paper, will be used to absorb moisture from the inside surface of the nostril. The special absorptive paper will be placed inside the nostril and left for a period of 2 minutes to absorb the nasal lining fluid before being removed, gently sucking up fluid like blotting paper. Putting the paper into the nose can tickle, and cause your eyes to water a little. However, the nasosorption does not hurt and our method has proved to be well tolerated in babies, children and adults. The paper absorbs the nasal fluid and many substances produced by the nasal cells can then be extracted from the paper and measured in the laboratory.
3. Nasal scrape (nasal curettage or Rhinoprobe): A small sterile disposable plastic probe will be inserted into the nose and will be gently pressed against the inside surface lining of the nostril. The 3 inch long probe has a tiny scoop on the end, which can barely be see. 24 tiny samples from each nostril (a pinhead, 2mm, of tissue) will be taken from a part of the nose that has a reduced nerve supply to limit any discomfort. Taking this sample does not cause bleeding, but may cause some mild discomfort, and may make the eyes water slightly. The probe will collect nasal cells from the surface of the nostril which will then be sent for analysis. This method has been performed on many adults, children, and babies, and has been very well tolerated.
4. Special Sampling Probe (SSP): The nasal surface lining fluid may also be collected using a special sampling probe or SSP that uses an electrospray to bounce droplets off the nasal lining fluid. This will be done by continuously sampling for a few hours from a single nostril. When using this special sampling probe (SSP) in people's noses, there is a slight tickling sensation while the sample is being taken. This can barely be noticed.

STATISTICAL ANALYSIS

The distribution of data will be assessed by the ShapiroWilks test, which determines whether the data has a normal (parametric) or non-normal (non-parametric) distribution.

Normal data will be displayed graphically as:

* arithmetic means and standard error of means (SEM)
* or means with SDs
* or means with confidence intervals (CIs)

Non-normal data will be displayed graphically as:

Box-whisker: median, quartiles, range

For non-normal data the differences from baseline will be measured for active challenge agent (at different doses) and placebo at each time point, and the AUC calculated. The differences in AUC from placebo (active placebo) are calculated, and the significance tested with the nonparametric Wilcoxon signed rank test(single population). Area under the curve (AUC) shall be sued over different defined times depending on the nasal challenge agent.

ELIGIBILITY:
INCLUSION CRITERIA

GENERAL FOR ALL SUBJECTS

* Males and females aged 18 to 60 years
* Current non-smokers for last year, maximum of 10 cigs per month, with a smoking history of <5 pack years
* Body mass index in the range18-39

HEALTHY NON-ATOPIC VOLUNTEERS

* Negative skin prick tests to a range of 6 common aeroallergens: cat, dog, grass pollen, tree pollen, house dust mite, fungal spores
* Normal blood eosinophil count.

ATOPIC SUBJECTS WITH TIMOTHY GRASS POLLEN SENSITIVITY

* A clinical history of seasonal grass pollen allergic rhinitis: sneezing, running and itching nose, nasal drip in the UK grass pollen summer season (May-July).
* Specific allergy confirmed by positive intra-epidermal skin prick test to Timothy grass pollen extract (Soluprick, Phleum pratense; ALK, Horsholm, Denmark), a positive reaction being a raised wheal of diameter >3mm larger than a negative saline control.

ASTHMATIC SUBJECTS WITH TIMOTHY GRASS POLLEN SENSITIVITY

* Seasonal grass pollen allergic rhinitis: sneezing, running and itching nose, nasal drip in the UK grass pollen summer season (May-July).
* Specific allergy confirmed by positive intra-epidermal skin prick test to Timothy grass pollen extract (Soluprick, Phleum pratense; ALK, Horsholm, Denmark), a positive reaction being a raised wheal of diameter >3mm larger than a negative saline control.
* Half the asthmatics have clinical history and diagnosis of asthma, requiring therapy with occasional inhaled beta-agonists, but no inhaled corticosteroids for the past 28 days. Half the asthmatics receive regular combined inhaled corticosteroids and long-acting beta-agonists (ICS/LABA)
* For those asthmatics in the resiquimod (TLR 7/8 agonist) arm:

Methacholine PC20 < 8mg/ml

SUBJECTS WITH LATENT TUBERCULOSIS

* Healthy with no lung nor systemic symptoms
* Positive blood Interferon-γ release assay (IGRA): Quantiferon TB Gold- in-Tube (QFT-it), >0.35 IU/ml IFN-γ versus control
* Tuberculin skin test (TST), using RT23 tuberculin purified protein derivative (PPD), from Statens Serum Institut (SSI) of Copenhagen. 2 tuberculin units (TU) in 0.1ml injected intradermally (id) : >6mm to <25mm of induration at 48-72h.
* Normal chest X-ray (CXR) or CT scan if performed routinely for clinical reasons

HEALTHY INTERFERON-γ RELEASE ASSAY (IGRA) NEGATIVE VOLUNTEERS

* Age and sex matched to latent TB subjects
* Healthy with no lung nor systemic symptoms
* Negative blood Interferon-γ release assay (IGRA): Quantiferon TB Gold- in-Tube (QFT-it), <0.35 IU/ml IFN-γ versus control
* Tuberculin skin test (TST), using RT23 tuberculin purified protein derivative (PPD), from Statens Serum Institut (SSI) of Copenhagen.
* 2 tuberculin units (TU) in 1ml injected intradermally (id): <6mm of induration at 48-72h.
* Chest X-ray is not required

EXCLUSION CRITERIA

GENERAL

* Recent infections in past 14 days before screening: especially upper respiratory tract illnesses (including colds and influenza), sore throats, sinusitis, infective conjunctivitis.
* Lower respiratory tract infection in past 28 days
* Signs or symptoms of significant nasal anatomical defects, hypertrophy of turbinates, major septum deviation, nasal polyposis injury, ulceration or recurrent sinusitis
* Previous nasal or sinus surgery
* Systemic illnesses that might affect nasal immune responses
* Medical therapy other than that permitted for contraception.
* Treatment with local or systemic corticosteroids during the previous 1 month
* Anti-inflammatory therapy: including non-steroidal anti-inflammatory drugs (NSAIDs)
* tuberculosis at any stage in life
* active infectious disease
* cardiovascular diseases
* respiratory (other than hay fever or asthma where specified)
* hepatic, gastrointestinal, renal, endocrine, infective, haematological, autoimmune, rheumatological, neurological, dermatological,
* neoplastic conditions
* metabolic diseases and extreme obesity
* depression and psychiatric disorders
* Non-smokers: up to 10 cigarettes a year is permitted
* Participation in a therapeutic drug trial in the prior 30 days.
* Inability or unwillingness to use contraception if the patient is a female of child-bearing age.
* Pregnant or breast feeding women
* Inability to provide informed consent

HEALTHY NON-ATOPIC VOLUNTEERS

* Clinical history of allergic rhinitis, allergic asthma or eczema

SUBJECTS WITH LATENT TUBERCULOSIS

* Clinical history of active symptomatic tuberculosis (TB) infection
* Chemoprophylaxis for TB

HEALTHY INTERFERON-γ RELEASE ASSAY (IGRA) NEGATIVE VOLUNTEERS

* Clinical history of TB infection
* Active nasal allergy
* BCG vaccination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Hansel, FRCPath, PhD, Principal Investigator — Imperial College London; Peter JM Openshaw, FRCP, PhD, FRSB, FMedSci, Study Director — Imperial College London; Robin Shattock, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Respiratory Research Unit (ICRRU), St Mary's Hospital, Paddington, London, United Kingdom

REFERENCES:
- [Background] Hansel TT, Johnston SL, Openshaw PJ. Microbes and mucosal immune responses in asthma. Lancet. 2013 Mar 9;381(9869):861-73. doi: 10.1016/S0140-6736(12)62202-8. PMID 23428115
- [Background] Chawes BL, Edwards MJ, Shamji B, Walker C, Nicholson GC, Tan AJ, Folsgaard NV, Bonnelykke K, Bisgaard H, Hansel TT. A novel method for assessing unchallenged levels of mediators in nasal epithelial lining fluid. J Allergy Clin Immunol. 2010 Jun;125(6):1387-1389.e3. doi: 10.1016/j.jaci.2010.01.039. Epub 2010 Mar 20. No abstract available. PMID 20304470
- [Background] Nicholson GC, Kariyawasam HH, Tan AJ, Hohlfeld JM, Quinn D, Walker C, Rodman D, Westwick J, Jurcevic S, Kon OM, Barnes PJ, Krug N, Hansel TT. The effects of an anti-IL-13 mAb on cytokine levels and nasal symptoms following nasal allergen challenge. J Allergy Clin Immunol. 2011 Oct;128(4):800-807.e9. doi: 10.1016/j.jaci.2011.05.013. Epub 2011 Jun 29. PMID 21719078
- [Background] Scadding GW, Calderon MA, Bellido V, Koed GK, Nielsen NC, Lund K, Togias A, Phippard D, Turka LA, Hansel TT, Durham SR, Wurtzen PA. Optimisation of grass pollen nasal allergen challenge for assessment of clinical and immunological outcomes. J Immunol Methods. 2012 Oct 31;384(1-2):25-32. doi: 10.1016/j.jim.2012.06.013. Epub 2012 Jun 30. PMID 22759401
- [Background] Ekman AK, Virtala R, Fransson M, Adner M, Benson M, Jansson L, Cardell LO. Systemic up-regulation of TLR4 causes lipopolysaccharide-induced augmentation of nasal cytokine release in allergic rhinitis. Int Arch Allergy Immunol. 2012;159(1):6-14. doi: 10.1159/000335196. Epub 2012 Apr 27. PMID 22555057
- [Background] Walrath JR, Silver RF. The alpha4beta1 integrin in localization of Mycobacterium tuberculosis-specific T helper type 1 cells to the human lung. Am J Respir Cell Mol Biol. 2011 Jul;45(1):24-30. doi: 10.1165/rcmb.2010-0241OC. Epub 2010 Aug 19. PMID 20724551
- [Background] Dhariwal J, Kitson J, Jones RE, Nicholson G, Tunstall T, Walton RP, Francombe G, Gilbert J, Tan AJ, Murdoch R, Kon OM, Openshaw PJ, Hansel TT. Nasal Lipopolysaccharide Challenge and Cytokine Measurement Reflects Innate Mucosal Immune Responsiveness. PLoS One. 2015 Sep 14;10(9):e0135363. doi: 10.1371/journal.pone.0135363. eCollection 2015. PMID 26367003

RESULTS

PARTICIPANT FLOW:
Groups:
- Poly ICLC Dose Escalation: Poly ICLC nasal challenge dose esalation: 10ug, 100ug, 500ug within same volunteers
- R848 High Dose: R848 nasal challenge with high dose 10ug
- Grass Pollen: Timothy Grass Pollen nasal challenge: Dose: 5000 SQ-U/100µl
- Vitamin D Supplementation: Vitamin D 4000U oraly daily
Period: Overall Study
Arm/Group | Poly ICLC Dose Escalation | Poly ICLC Highest Dose | Poly I:C Single Dose | R848 High Dose | R848 Low Dose | Grass Pollen | Vitamin D Supplementation | Tuberculin
Started | 8 | 4 | 4 | 9 | 35 | 15 | 16 | 2
Completed | 8 | 4 | 4 | 9 | 35 | 15 | 16 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Poly ICLC Dose Escalation: Dose esalation within same volunteers: 10ug, 100ug, 500ug
- Poly ICLC Highest Dose: Single dose: 1000ug
- Poly I:C Single Dose: Poly I:C nasal challenge single dose: 500ug
- R848 High Dose: R848 nasal challenge high dose: 10ug
- R848 Low Dose: R848 nasal challenge low dose: 1-2ug (0.02ug/kg)
- Grass Pollen: Timothy Grass Pollen nasal challenge: 5000 SQ-U/100µl
- Total: Total of all reporting groups
Arm/Group | Poly ICLC Dose Escalation | Poly ICLC Highest Dose | Poly I:C Single Dose | R848 High Dose | R848 Low Dose | Grass Pollen | Vitamin D Supplementation | Tuberculin | Total
Number analyzed (Participants) | 8 | 4 | 4 | 9 | 35 | 15 | 16 | 2 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 4 | 9 | 35 | 15 | 16 | 2 | 93
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 8 | 20 | 7 | 8 | 1 | 54
  Male | 4 | 1 | 1 | 1 | 15 | 8 | 8 | 1 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: IFN-y Protein Response in Mucosal Lining Fluid
Description: The primary outcome measure is IFN-y in nasal mucosal lining fluid after nasal challenge
Time Frame: 0, 1, 2, 3, 4, 6, 8 hours post-dose
Measure: Mean (95% Confidence Interval); unit: pg/hr/ml
Groups:
- Poly ICLC Dose Escalation: Poly ICLC nasal challenge dose escalation: 10ug, 100ug, 500ug
- Poly ICLC High Dose: Poly ICLC nasal challenge single dose of 1000ug
- Poly I:C Single Dose: Poly I:C nasal challenge 500ug
Arm/Group | Poly ICLC Dose Escalation | Poly ICLC High Dose | Poly I:C Single Dose | R848 High Dose | R848 Low Dose | Grass Pollen | Vitamin D Supplementation | Tuberculin
Number analyzed (Participants) | 8 | 4 | 4 | 9 | 35 | 15 | 16 | 2
pg/hr/ml | NA [NA to NA] — Below the level of detection | 3.29 [1.84 to 4.74] | 9.42 [4.76 to 14.08] | 8.20 [6.30 to 10.11] | 5.10 [3.88 to 6.32] | NA [NA to NA] — Below the level of detection | NA [NA to NA] — Below the level of detection | NA [NA to NA] — Insufficient number of participants. Samples were therefore not assessed for cytokine measurements.

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Poly ICLC Higest Dose: Poly ICLC nasal challenge 1000ug
- R848 High Dose: R848 high dose 10ug
- R848 Low Dose: R848 low dose 1-2ug 0.02ug/kg
Arm/Group | Poly ICLC Dose Escalation | Poly ICLC Higest Dose | Poly I:C Single Dose | R848 High Dose | R848 Low Dose | Grass Pollen | Vitamin D Supplementation | Tuberculin
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/4 | 0/9 | 0/35 | 0/15 | 0/16 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/4 | 0/9 | 0/35 | 0/15 | 0/16 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/4 | 4/9 | 11/35 | 0/15 | 0/16 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly ICLC Dose Escalation (N=8) | Poly ICLC Higest Dose (N=4) | Poly I:C Single Dose (N=4) | R848 High Dose (N=9) | R848 Low Dose (N=35) | Grass Pollen (N=15) | Vitamin D Supplementation (N=16) | Tuberculin (N=2)
Fever (Immune system disorders) | 0 | 0 | 0 | 3 (3) | 0 | 0 | 0 | 0 — Fever >37.2 C
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 (3) | 3 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 (3) | 1 | 0 | 0 | 0
Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 (3) | 6 | 0 | 0 | 0
Blocked nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 11 | 0 | 0 | 0 — Blocked nose/rhinitis

LIMITATIONS AND CAVEATS:
Tuberculin nasal challenge did not proceed to full enrollment due to insufficient numbers of eligible participants. Samples were therefore not assessed for cytokine measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02090374/Prot_SAP_000.pdf